CLINICAL TRIAL: NCT06744972
Title: Native Tissue Repair in Pelvic Organ Prolapse -Long-term Results and Risk of Re-operation
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pia Heinonen, MD, PhD, head of section, gynaecology, Turku University Hospital
Other Study IDs: T43/2016
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Organ Prolapse; Cystocele
Keywords: Recurrence; Native tissue repair
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the recurrence of pelvic organ prolapse and the rate of re-operation after primary surgery for anterior vaginal wall prolapse with native tissue repair in long term follow-up.

DETAILED DESCRIPTION:
This was a retrospective cohort study including patients undergoing their first surgical intervention for pelvic organ prolapse in Turku University Hospital gynecology department in the years 2000-2005. The point of interest was to study patients with prolapse of the anterior vaginal compartment (i.e. cystocele) with native tissue repair surgical approach as treatment. We made a search from the medical database of surgical procedures for operation codes LEF00 (i.e.anterior colporraphy and LEF13 (i.e. vaginal hysterectomy of descended uterus with/without vaginal/perineal molding) during the studied period. Initially, we found 699 patients with matching operating codes and for those, we went through their medical records. From the final study population, we excluded those who had previously had an operation for pelvic organ prolapse and those whose primary operation didn't include anterior colporraphy and those who weren't eligible for long term follow-up. Thus, the study population constituted of 392 subjects who were followed through medical records until the end of October 2018.

From the medical records, we collected the day of birth, the date of the primary operation, body mass index, history of vaginal childbirth and cesarean section (if available), history of incontinence surgery, the grade of cystocele and diagnosis and before surgery, the operation code and executed surgical procedures, possible complications, and the history of possible re-operations. Also, the date of death was reported as well as the date of changing residence outside the Hospital District of Varsinais-Suomi.

All gathered information were saved without personal details.

ELIGIBILITY:
Inclusion Criteria:

* cystocele treated with native tissue surgery, medical records reaching until the end of follow-up period

Exclusion Criteria:

* history of previous pelvic organ prolapse surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients treated for cystocele for the first time with native tissue repair.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Rate of re-operations | Long-term, at least 5 years follow up.
  Evaluate the risk of re-operation for pelvic organ prolapse and recurrence of surgically treated cystocele.

IPD SHARING:
Plan to Share IPD: No